CLINICAL TRIAL: NCT01511809
Title: Efficacy of Atazanavir / Ritonavir Monotherapy as Maintenance in Patients With Viral Suppression. Randomized, Open Label Non Inferiority Trial. A Phase 3 Study.
Brief Title: Efficacy of Atazanavir/Ritonavir Monotherapy as Maintenance in Patients With Viral Suppression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Castagna Antonella, Co- Investigator, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MODAt
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: HIV-1 Infection
Keywords: HIV-1
MeSH Terms: interventions — Atazanavir Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atazanavir/ritonavir monotherapy (Experimental): Patients will simplify therapy to ATV/RTV 300mg/100mg OD as monotherapy
  Interventions: Drug: Atazanavir/ritonavir monotherapy
- Atazanavir/ritonavir triple therapy (No Intervention): Patients will continue the same regimen ATV/RTV 300mg/100mg OD plus 2 NRTIs as backbone

INTERVENTIONS:
Drug: Atazanavir/ritonavir monotherapy — Monotherapy Simplification Strategy with Atazanavir/ritonavir 300/100 mg once daily for 96 weeks.
  Other Names: ATV/r monotherapy
  Arms: Atazanavir/ritonavir monotherapy

SUMMARY:
The study will assess whether Atazanavir/ritonavir monotherapy provides a non-inferior proportion of virological efficacy with respect to ATV/RTV + 2 NRTIs in patients with stable suppressed viremia and no prior virologic failures.

DETAILED DESCRIPTION:
This is a randomised (1:1), multicentre, comparative, parallel-group, prospective, open label, non-inferiority controlled clinical trial.

Enrolled patients, taking an ATV/r based HAART and with stable HIV-RNA < 50c/ml (24 weeks), will be randomized to:

* continue the same regimen ATV/RTV 300mg/100mg OD plus 2 NRTIs (according to the specific dosing schedule) as backbone (HAART arm) with ATV/r
* or simplify therapy to ATV/RTV 300mg/100mg OD as monotherapy (Monotherapy arm) with ATV/r The study follow up will be 96 weeks after randomization and primary objective will be evaluated at week 48.

Patients will be followed every 4 weeks for the first 16 weeks, and then every 8 weeks until week 48, then every 12 weeks until week 96 or discontinuation ; at each visit the following evaluations will be performed:

* clinical assessment.
* routine laboratory tests (hematological tests and hematochemistry) including creatinine, phosphorus, calcium, alkaline phosphatase, gammaGT; urine analysis, lipid profile, level of HIV-RNA and CD4 cell counts.

During follow-up, at randomization, week 48, week 96 or discontinuation, patients will additionally undergo:

* Fat redistribution evaluation by DEXA (dual-energy X-ray absorptiometry
* Vertebral and femoral bone mineral density evaluation by DEXA.
* ECG;
* Glicate haemoglobin.
* Adherence assessment (questionnaire and/or pills counts).
* Neurocognitive evaluation [HIV-associated neurocognitive disorders (HANDs) evaluated by validated neuropsychological tests].

In case of viral rebound (defined as 2 consecutive measurement of HIV-RNA > 50 c/ml) patients will be immediately contacted in order to perform genotypic tests. Furthermore a plasma PK analysis will also be performed. Any patients with virological rebound will be selected for a reintensification therapy with NRTIs and if not suppressed after 12 weeks they will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients
* age > 18 years
* On treatment with ATV/r plus 2 NRTIs for at least 48 weeks
* Virological suppression (HIV-RNA<50 c/ml) by at least 24 weeks with ATV/r plus 2 NRTIs
* No virologic failure after the initiation of the first antiretroviral therapy. Previous treatment changes due to toxicity or treatment simplifications will be permitted only if occurred with documented virological suppression.
* CD4 cells nadir >100 cells/µL
* PPI and H2-receptor antagonists as follows: the proton-pump inhibitors should not be used; if H2-receptor antagonists are co-administered, a dose equivalent to famotidine 20 mg BID should not be exceeded.

Exclusion Criteria:

* Pregnancy and breast feeding women
* AIDS defining events
* Evidence of active HBV infection (HBsAg positive)
* Previous virological failure
* History of resistance to ATV
* Use of contraindicated medications

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Lazzarin, Professor, Principal Investigator — Ospedale San Raffaele
Locations (1):
- Infectious Diseases Department Fondazione Centro San Raffaele, Milan, Lombardy, Italy

REFERENCES:
- [Background] Delfraissy JF, Flandre P, Delaugerre C, Ghosn J, Horban A, Girard PM, Norton M, Rouzioux C, Taburet AM, Cohen-Codar I, Van PN, Chauvin JP. Lopinavir/ritonavir monotherapy or plus zidovudine and lamivudine in antiretroviral-naive HIV-infected patients. AIDS. 2008 Jan 30;22(3):385-93. doi: 10.1097/QAD.0b013e3282f3f16d. PMID 18195565
- [Background] Cameron DW, da Silva BA, Arribas JR, Myers RA, Bellos NC, Gilmore N, King MS, Bernstein BM, Brun SC, Hanna GJ. A 96-week comparison of lopinavir-ritonavir combination therapy followed by lopinavir-ritonavir monotherapy versus efavirenz combination therapy. J Infect Dis. 2008 Jul 15;198(2):234-40. doi: 10.1086/589622. PMID 18540803
- [Background] Pulido F, Arribas JR, Delgado R, Cabrero E, Gonzalez-Garcia J, Perez-Elias MJ, Arranz A, Portilla J, Pasquau J, Iribarren JA, Rubio R, Norton M; OK04 Study Group. Lopinavir-ritonavir monotherapy versus lopinavir-ritonavir and two nucleosides for maintenance therapy of HIV. AIDS. 2008 Jan 11;22(2):F1-9. doi: 10.1097/QAD.0b013e3282f4243b. PMID 18097218
- [Background] Arribas JR, Delgado R, Arranz A, Munoz R, Portilla J, Pasquau J, Perez-Elias MJ, Iribarren JA, Rubio R, Ocampo A, Sanchez-Conde M, Knobel H, Arazo P, Sanz J, Lopez-Aldeguer J, Montes ML, Pulido F; OK04 Study Group. Lopinavir-ritonavir monotherapy versus lopinavir-ritonavir and 2 nucleosides for maintenance therapy of HIV: 96-week analysis. J Acquir Immune Defic Syndr. 2009 Jun 1;51(2):147-52. doi: 10.1097/QAI.0b013e3181a56de5. PMID 19349870
- [Background] Arribas JR, Horban A, Gerstoft J, Fatkenheuer G, Nelson M, Clumeck N, Pulido F, Hill A, van Delft Y, Stark T, Moecklinghoff C. The MONET trial: darunavir/ritonavir with or without nucleoside analogues, for patients with HIV RNA below 50 copies/ml. AIDS. 2010 Jan 16;24(2):223-30. doi: 10.1097/QAD.0b013e3283348944. PMID 20010070
- [Background] Katlama C, Valantin MA, Algarte-Genin M, Duvivier C, Lambert-Niclot S, Girard PM, Molina JM, Hoen B, Pakianather S, Peytavin G, Marcelin AG, Flandre P. Efficacy of darunavir/ritonavir maintenance monotherapy in patients with HIV-1 viral suppression: a randomized open-label, noninferiority trial, MONOI-ANRS 136. AIDS. 2010 Sep 24;24(15):2365-74. doi: 10.1097/QAD.0b013e32833dec20. PMID 20802297
- [Background] Swindells S, DiRienzo AG, Wilkin T, Fletcher CV, Margolis DM, Thal GD, Godfrey C, Bastow B, Ray MG, Wang H, Coombs RW, McKinnon J, Mellors JW; AIDS Clinical Trials Group 5201 Study Team. Regimen simplification to atazanavir-ritonavir alone as maintenance antiretroviral therapy after sustained virologic suppression. JAMA. 2006 Aug 16;296(7):806-14. doi: 10.1001/jama.296.7.806. PMID 16905786
- [Background] Karlstrom O, Josephson F, Sonnerborg A. Early virologic rebound in a pilot trial of ritonavir-boosted atazanavir as maintenance monotherapy. J Acquir Immune Defic Syndr. 2007 Apr 1;44(4):417-22. doi: 10.1097/QAI.0b013e31802e2940. PMID 17159658
- [Background] Wilkin TJ, McKinnon JE, DiRienzo AG, Mollan K, Fletcher CV, Margolis DM, Bastow B, Thal G, Woodward W, Godfrey C, Wiegand A, Maldarelli F, Palmer S, Coffin JM, Mellors JW, Swindells S. Regimen simplification to atazanavir-ritonavir alone as maintenance antiretroviral therapy: final 48-week clinical and virologic outcomes. J Infect Dis. 2009 Mar 15;199(6):866-71. doi: 10.1086/597119. PMID 19191590
- [Background] Vernazza P, Daneel S, Schiffer V, Decosterd L, Fierz W, Klimkait T, Hoffmann M, Hirschel B. The role of compartment penetration in PI-monotherapy: the Atazanavir-Ritonavir Monomaintenance (ATARITMO) Trial. AIDS. 2007 Jun 19;21(10):1309-15. doi: 10.1097/QAD.0b013e32814e6b1c. PMID 17545707

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atazanavir/Ritonavir Monotherapy | Atazanavir/Ritonavir Triple Therapy
Started | 58 | 59
Completed | 51 | 52
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atazanavir/Ritonavir Monotherapy | Atazanavir/Ritonavir Triple Therapy | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 41.4 [35.4 to 47.7] | 41.7 [36.6 to 49.8] | 41.5 [35.6 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 42 | 45 | 87
Region of Enrollment [Number; unit: participants]
  Italy | 51 | 52 | 103
nadir CD4+ [Median (Inter-Quartile Range); unit: cells/mm3] — Lowest CD4+ value among those recorded since the first HIV positive test up to the start of MODAt study
  cells/mm3 | 274 [221 to 355] | 278 [183 to 364] | 276 [211 to 361]
Years of antiretroviral treatment [Median (Inter-Quartile Range); unit: years] | 25 [16 to 47] | 25 [18 to 54] | 25 [17 to 53]
HIV-1 RNA <50 copies/ml [Median (Inter-Quartile Range); unit: months] — Quantitative value of HIV-1 RNA copies/ml in plasma. HIV-1 RNA below 50 copies/ml (detection limit) is an indicator of efficacy of the antiretroviral therapy
  months | 20 [10 to 49] | 18 [12 to 49] | 19 [11 to 49]
HIV-RNA at ARV start [Median (Inter-Quartile Range); unit: copies/mL] | 79399 [31046 to 183613] | 42630 [9696 to 123700] | 59062 [10834 to 165850]
CD4+ [Median (Inter-Quartile Range); unit: cells/mm3] | 599 [457 to 774] | 570 [417 to 735] | 575 [432 to 744]
HCV coinfection [Number; unit: participants]
  Present | 11 | 10 | 21
  Absent | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Treatment Failure (TF)
Description: Proportion of patients with treatment failure defined as having one of the following events: confirmed viral rebound (CVR) or treatment discontinuation for any cause. CVR was established when 2 consecutive viral load values (HIV-1 RNA)>50 copies/mL occurred within 2 weeks during follow-up. In case of CVR, patients treated with atazanavir/ritonavir monotherapy had to re-introduce their previous 2NRTIs (re-intensification) and, if not suppressed (HIV-1 RNA <50 copies /ml) after 12 weeks, discontinued from the study. Re-intensification was considered as treatment failure in the primary analysis conducted according to the intention-to-treat principle (intention-to-treat analysis with re-intensification equal failure, ITT=Failure) while it was not in the secondary analysis (intention-to-treat analysis with re-intensification equal success, ITT=Success).
Time Frame: Up to week 48
Measure: Number; unit: percentage of patients
Arm/Group | Atazanavir/Ritonavir Monotherapy | Atazanavir/Ritonavir Triple Therapy
Number analyzed (Participants) | 51 | 52
percentage of patients
  ITT=Failure analysis | 27.5 | 15.4
  ITT=Success analysis | 7.9 | 15.4
Statistical Analysis 1: Comparison: Atazanavir/Ritonavir Monotherapy vs Atazanavir/Ritonavir Triple Therapy; Here are reported the results of the 48-week interim analyses according to the intention-to-treat (ITT) principle. ITT=F (with re-intensification=failure) and the ITT=S (with re-intensification=success) treatment failure results are shown. Based on the efficacy data review, in June 2013, an independent Data and Safety Monitoring Board (DSMB) recommended to stop further patients' enrolment and to follow-up the enrolled patients until 96 weeks, after having signed an updated informed consent; Test type: Non-Inferiority or Equivalence — A lower limit of the 95% confidence interval of the difference between the two proportions of treatment failure (triple therapy-monotherapy) below the pre-specified margin of non-inferiority of -10% established inferiority. A sample size of 342 patients (171 per treatment arm) provided 80% power (one-sided, alpha 0.05) to establish non-inferiority of ATV/r monotherapy as compared to ATV/r triple therapy with an overall treatment failure (TF) rate of 15% at week 48; difference between TF proportions = 15

2. Secondary Outcome: Efficacy and Safety
Description: Proportion of pts with confirmed virological and treatment failure at w96. Change in CD4 cell counts.
  Occurrence of viral resistance to atazanavir in pts with confirmed virologic failure.
  Proportion of pts with adverse events, with ≥grade 2 adverse events or abnormal laboratory tests, proportion of pts with side effects leading to discontinuation.
  Body fat redistribution and vertebral and femoral bone mineral density. Adherence changes; changes in HIV-associated neurocognitive disorders. Difference in levels of activated Tcells and pro-inflammatory cytokines between treatment groups.
Time Frame: week 96
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to week 48
Arm/Group | Atazanavir/Ritonavir Monotherapy | Atazanavir/Ritonavir Triple Therapy
Serious Adverse Events (participants affected / at risk) | 2/51 | 0/52
Other Adverse Events (participants affected / at risk) | 1/51 | 7/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atazanavir/Ritonavir Monotherapy (N=51) | Atazanavir/Ritonavir Triple Therapy (N=52)
acute coronary stenosis (Cardiac disorders) | 1 | 0
left basal pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atazanavir/Ritonavir Monotherapy (N=51) | Atazanavir/Ritonavir Triple Therapy (N=52)
acute hepatitis (Hepatobiliary disorders) | 1 | 1
nephrolitiasis (Renal and urinary disorders) | 0 | 2
cholecystitis due to cholelithiasis (Hepatobiliary disorders) | 0 | 1
hyperuricemia (Renal and urinary disorders) | 0 | 1
gross haematuria with proteinuria (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No